CLINICAL TRIAL: NCT04594044
Title: Group Therapy Versus Individual Therapy in Children and Adolescents With Tourette Syndrome and Chronic Tic Disorder
Brief Title: Group Therapy Versus Individual Therapy for Tourette Syndrome and Chronic Tic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Judith Becker Nissen, MD, PhD, senior researcher, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-72-216-15
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2020-10

CONDITIONS: Chronic Tic Disorder
Keywords: Habit reversal training; Exposure response prevention; Children and adolescents
MeSH Terms: conditions — Tic Disorders

STUDY DESIGN:
Intervention Model Description: In an open randomized controlled study, youth were randomized to either individualized, or group treatment. Both therapies included nine sessions, and the parents were offered one group-session. Treatment effect was evaluated after 8 and 9 months, and after one year of follow-up
Who Masked: Outcomes Assessor
Masking Description: Evaluations of treatment response were made by an independent evaluator who was not blinded to the treatment allocation, yet not involved in the treatment of the patient, and blinded to any previous evaluations. The evaluators were a specialized psychologist and a child and adolescent psychiatrist with several years of experience in diagnosing, evaluating and treating tic disorders. A random sample of 10% were audiotaped and evaluated by another rater with extensive experience and expertise in the use of the YGTSS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual HRT and ERP (Experimental): Individual treatment with habit reversal training (HRT) and exposure response prevention (ERP) according to a protocol
  Interventions: Behavioral: tics training including habit reversal training and exposure response prevention
- Group HRT and ERP (Experimental): Group treatment with habit reversal training (HRT) and exposure response prevention (ERP) according to a protocol
  Interventions: Behavioral: tics training including habit reversal training and exposure response prevention

INTERVENTIONS:
Behavioral: tics training including habit reversal training and exposure response prevention — In an open randomized controlled study, youth were randomized to either individualized, or group treatment. Both therapies included nine sessions, and the parents were offered one group-session.

SUMMARY:
Chronic tic disorder (CTD) may have a huge impact on life quality. Habit Reversal Training (HRT) and Exposure Response Prevention (ERP) are effective therapeutic modalities. This study examined the effect of a combined treatment using both HRT and ERP in children and adolescents with CTD. The treatment outcome was examined as an individual treatment compared to a group setting. There was no control group. The study examined both acute outcome and outcome at one year of follow-up. Predictive factors for treatment outcome were evaluated.

DETAILED DESCRIPTION:
Chronic tic disorder (CTD) may have a huge impact on life quality. Habit Reversal Training (HRT) and Exposure Response Prevention (ERP) are known to be effective therapeutic modalities. Little is known about the effect of group therapy, the effect of combining HRT and ERP training, and of the long-term effect of treatment. This study therefore wanted to examine the effect of a combined treatment using both HRT and ERP in children and adolescents with CTD. The participants were randomized to treatment either in groups or in an individual setting. The parents were included in the training programme. The participants were asked to fulfill questionnaires concerning anxiety, mood, life quality, their thoughts about tics and the experienced premonitory urge. Furthermore, they were interviewed with the semistructured interview Yale Global Tic Severity Scale (YGTSS).

Data was obtained from patient files as to examine possible predictors of both acute and long-term treatment effects. The evaluators were a specialized psychologist and a child and adolescent psychiatrist with several years of experience in diagnosing, evaluating and treating tic disorders. A random sample of 10% were audiotaped and evaluated by another rater with extensive experience and expertise in the use of the YGTSS. The evaluator was not blinded to the treatment allocation, yet not involved in the treatment of the patient, and blinded to any previous evaluations

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of either Tourette syndrome or a chronic motor/vocal tics disorder
* Moderate or greater severity corresponding to a total score on the Yale Global Tic Severity Scale (YGTSS) higher than 13 (higher than nine if only motor or vocal tics were described)

Exclusion Criteria:

1. Disorders that required immediate treatment

   * psychotic disorder
   * primary severe depression
   * suicidal ideation or attempts
   * primary severe anorexia nervosa
2. Disorders that makes participation difficult

   * IQ below 70
   * a life-time diagnosis of pervasive developmental disorder
3. Treatment with HRT or ERP during the last six months.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change of baseline Yale Global Tic Severity Scale (YGTSS) at 16 weeks, 24 weeks, 40 weeks and 68 weeks | Baseline,16 weeks, 24 weeks, 40 weeks, 68 weeks
  Measures the change in Total tic score and functional impairment at different end points on the Yale Global Tic Severity Scale (unabbreviated scale title). Interval 0-100, high score means a worse outcome

SECONDARY OUTCOMES:
Change of baseline Premonitory urge (PUTS) at 6 weeks, 16 weeks, 24 weeks, and 68 weeks | Baseline, 6 weeks, 16 weeks, 24 weeks, 68 weeks
  Measures the change of baseline premonitory urge score at different end points on the Premonitory Urge scale (unabbreviated scale title). Interval 1-4, high score means a worse outcome
Change of baseline Beliefs About Tics Scale (BATS) at 6 weeks, 16 weeks, 24 weeks, and 68 weeks | Baseline, 6 weeks, 16 weeks, 24 weeks, 68 weeks
  Measures the change of baseline Beliefs About Tics Scale score at different end points on the Beliefs About Tics Scale (unabbreviated scale title). Interval 1-4, high score means a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Judith Nissen, Principal Investigator — Department of Child and Adolescent Psychiatry, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
In accordance to Danish law, personal data cannot be shared

REFERENCES:
- [Derived] Nissen JB, Carlsen AH, Thomsen PH. One-year outcome of manualised behavior therapy of chronic tic disorders in children and adolescents. Child Adolesc Psychiatry Ment Health. 2021 Feb 20;15(1):9. doi: 10.1186/s13034-021-00362-w. PMID 33610169